CLINICAL TRIAL: NCT00300755
Title: A Multicenter, Randomized, Double-Blind Study of the Clinical Outcomes, Safety and Tolerability of Multiple Doses of Pantoprazole Sodium Enteric-Coated Spheroids in Children Ages 1 to 5 With Endoscopically Proven Symptomatic Gastroesophageal Reflux Disease (GERD)
Brief Title: Study Evaluating Pantoprazole in Children With Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Nycomed (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3001B3-328
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Results first posted 2010-05-19 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Gastroesophageal Reflux
Keywords: GERD; Children; Child; Child, Preschool
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Arm 1- Low Dose pantoprazole
  Interventions: Drug: pantoprazole sodium enteric-coated spheroid
- 2 (Active Comparator): Arm 2- Medium Dose pantoprazole
  Interventions: Drug: pantoprazole sodium enteric-coated spheroid
- 3 (Active Comparator): Arm 3- High Dose pantoprazole
  Interventions: Drug: pantoprazole sodium enteric-coated spheroid

INTERVENTIONS:
Drug: pantoprazole sodium enteric-coated spheroid — pediatric spheroids taken daily x 8 weeks

SUMMARY:
To evaluate the clinical outcomes of treatment with oral pantoprazole in children 1 through 5 years of age with endoscopically proven symptomatic GERD.

ELIGIBILITY:
Inclusion Criteria:

* Ability to undergo endoscopy with required biopsy
* Ages 1 through 5 years
* Endoscopically confirmed GERD by positive endoscopic evidence of reflux related esophagitis or positive histologic evidence of esophagitis consistent with GERD Other inclusions apply.

Exclusion Criteria:

* History or presence of upper gastrointestinal anatomic or motor disorders
* Known current or active cow's milk allergy
* Malignancy
* Other exclusions apply.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (41):
- United States (35):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Oakland, California
  - Orange, California
  - Sacramento, California
  - San Diego, California
  - Wilmington, Delaware
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Peoria, Illinois
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Flint, Michigan
  - Southfield, Michigan
  - Jackson, Mississippi
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Egg Harbor, New Jersey
  - Morristown, New Jersey
  - Buffalo, New York
  - New York, New York
  - Oklahoma City, Oklahoma
  - Danville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Temple, Texas
  - Norfolk, Virginia
  - Charleston, West Virginia
  - Huntington, West Virginia
  - Milwaukee, Wisconsin
- Canada (6):
  - Edmonton, Alberta
  - St. John's, Newfoundland and Labrador
  - Hamilton, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Montreal, Quebec

REFERENCES:
- [Derived] Baker R, Tsou VM, Tung J, Baker SS, Li H, Wang W, Rath N, Maguire MK, Comer GM. Clinical results from a randomized, double-blind, dose-ranging study of pantoprazole in children aged 1 through 5 years with symptomatic histologic or erosive esophagitis. Clin Pediatr (Phila). 2010 Sep;49(9):852-65. doi: 10.1177/0009922810369253. Epub 2010 Jun 3. PMID 20522615

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the United States and Canada from May 2006 to February 2008.
Pre-assignment Details: Patients were screened for up to four weeks.
Groups:
- Low Dose Pantoprazole (Approximately 0.3 mg/kg): Capsules containing pantoprazole sodium-enteric coated spheroids (granules) 5 mg once daily for 8 weeks
- Medium Dose Pantoprazole (Approximately 0.6 mg/kg): Capsules containing pantoprazole sodium-enteric coated spheroids (granules) 10 mg once daily for 8 weeks
- High Dose Pantoprazole (Approximately 1.2 mg/kg): Capsules containing pantoprazole sodium-enteric coated spheroids (granules) 15 mg once daily for 8 weeks for patients ≥1 to <2 years. Capsules containing pantoprazole sodium-enteric coated spheroids (granules) 20 mg once daily for 8 weeks for patients from ≥2 to <6 years.
Period: Overall Study
Arm/Group | Low Dose Pantoprazole (Approximately 0.3 mg/kg) | Medium Dose Pantoprazole (Approximately 0.6 mg/kg) | High Dose Pantoprazole (Approximately 1.2 mg/kg)
Started | 18 | 21 | 21
Completed | 17 | 17 | 19
Not Completed | 1 | 4 | 2
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Pantoprazole (Approximately 0.3 mg/kg) | Medium Dose Pantoprazole (Approximately 0.6 mg/kg) | High Dose Pantoprazole (Approximately 1.2 mg/kg) | Total
Number analyzed (Participants) | 18 | 21 | 21 | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 2.67 (1.61) | 1.90 (1.18) | 2.76 (1.34) | 2.43 (1.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 13 | 23.0
  Male | 12 | 17 | 8 | 37.0

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Gastroesophageal Reflux Disease (GERD) Symptom Scores (WGSS)
Description: WGSS is the sum of 5 selected individual weekly GERD mean frequency scores: vomiting/regurgitation, choking/gagging, refusal to eat, difficulty swallowing and abdominal/belly pain. Symptoms were assessed using a parent-administered questionnaire. The score for each individual symptom ranged from 0 (no symptoms) to 3 (highest frequency of symptoms), giving a WGSS range of 0-15. Change = score at week of assessment minus baseline score. Final week was defined as the last 7 days of symptom scores collected in the treatment period.
Time Frame: Baseline and 8 weeks
Population: The primary efficacy population (mITT NERD) included all patients who were randomized and received ≥1 dose of test article and had nonerosive gastroesophageal reflux disease. Last observation carried forward (except for baseline data, which were not carried forward into the treatment period).
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Low Dose Pantoprazole (Approximately 0.3 mg/kg) | Medium Dose Pantoprazole (Approximately 0.6 mg/kg) | High Dose Pantoprazole (Approximately 1.2 mg/kg)
Number analyzed (Participants) | 18 | 19 | 19
units on scale
  Week 1 Change from Baseline | -0.89 (1.41) | 0.02 (0.99) | -0.47 (1.25)
  Week 2 Change from Baseline | -1.11 (1.29) | -0.11 (1.06) | -1.24 (1.42)
  Week 3 Change from Baseline | -1.31 (1.43) | -0.16 (1.23) | -1.38 (1.47)
  Week 4 Change from Baseline | -1.84 (1.95) | -0.20 (1.29) | -1.32 (1.36)
  Week 5 Change from Baseline | -2.05 (2.08) | -0.48 (1.31) | -1.30 (1.63)
  Week 6 Change from Baseline | -1.99 (1.83) | -0.61 (1.31) | -1.42 (1.59)
  Week 7 Change from Baseline | -2.44 (1.75) | -0.58 (1.38) | -1.58 (1.62)
  Week 8 Change from Baseline | -2.34 (1.81) | -0.60 (1.49) | -1.61 (1.61)
  Final Week Change from Baseline | -2.37 (1.74) | -0.64 (1.40) | -1.66 (1.64)
Statistical Analysis 1: Comparison: Low Dose Pantoprazole (Approximately 0.3 mg/kg); Within group analysis of final week change from baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Medium Dose Pantoprazole (Approximately 0.6 mg/kg); Within group analysis of final week change from baseline; Test type: Superiority or Other; p = 0.063, t-test, 2 sided
Statistical Analysis 3: Comparison: High Dose Pantoprazole (Approximately 1.2 mg/kg); Within group analysis of final week change from baseline; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: Low Dose Pantoprazole (Approximately 0.3 mg/kg) vs Medium Dose Pantoprazole (Approximately 0.6 mg/kg); Between group analysis of final week change from baseline; Test type: Superiority or Other; p = 0.004, ANCOVA; Analysis with treatment group and baseline age as fixed effects, and baseline GERD symptom score and baseline antacid use as covariates
Statistical Analysis 5: Comparison: Low Dose Pantoprazole (Approximately 0.3 mg/kg) vs High Dose Pantoprazole (Approximately 1.2 mg/kg); Between group analysis of final week change from baseline; Test type: Superiority or Other; p = 0.082, ANCOVA; [statistical method as in outcome 1, analysis 4]
Statistical Analysis 6: Comparison: Medium Dose Pantoprazole (Approximately 0.6 mg/kg) vs High Dose Pantoprazole (Approximately 1.2 mg/kg); Between group analysis of final week change from baseline; Test type: Superiority or Other; p = 0.217, ANCOVA; [statistical method as in outcome 1, analysis 4]

2. Secondary Outcome: Change in Individual Weekly Mean Frequency Score for Each Gastroesophageal Reflux Disease (GERD) Symptom Score From Baseline to Final Week
Description: Selected symptoms of GERD were assessed using a parent-administered questionnaire. The score for each symptom ranged from 0 (no symptom) to 3 (highest frequency of symptom), The weekly mean score was the sum of daily scores that week, divided by the number of days with scores for that week. Change = final week score minus baseline score. Final week was defined as the last 7 days of scores collected in the treatment period.
Time Frame: Baseline and 8 weeks
Population: The analysis population is all patients who were randomized and received ≥1 dose of test article and had nonerosive gastroesophageal reflux disease.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Low Dose Pantoprazole (Approximately 0.3 mg/kg) | Medium Dose Pantoprazole (Approximately 0.6 mg/kg) | High Dose Pantoprazole (Approximately 1.2 mg/kg)
Number analyzed (Participants) | 18 | 19 | 19
units on scale
  Vomiting/regurgitation | -0.77 (0.89) | -0.06 (0.28) | -0.25 (0.48)
  Choking/gagging | -0.43 (0.33) | -0.05 (0.48) | -0.47 (0.59)
  Refusal to eat | -0.34 (0.49) | -0.16 (0.61) | -0.26 (0.69)
  Difficulty swallowing | -0.42 (0.52) | -0.13 (0.49) | -0.39 (0.79)
  Abdominal/belly pain | -0.42 (0.49) | -0.24 (0.44) | -0.28 (0.49)
Statistical Analysis 1: Comparison: Low Dose Pantoprazole (Approximately 0.3 mg/kg); Within group analysis of final week change from baseline for symptom Vomiting/regurgitation; Test type: Superiority or Other; p = 0.002, t-test, 2 sided
Statistical Analysis 2: Comparison: High Dose Pantoprazole (Approximately 1.2 mg/kg); Within group analysis of final week change from baseline for symptom Vomiting/regurgitation; Test type: Superiority or Other; p = 0.033, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Dose Pantoprazole (Approximately 0.3 mg/kg); Within group analysis of final week change from baseline for symptom Choking/gagging; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 4: Comparison: High Dose Pantoprazole (Approximately 1.2 mg/kg); Within group analysis of final week change from baseline for symptom Choking/gagging; Test type: Superiority or Other; p = 0.002, t-test, 2 sided
Statistical Analysis 5: Comparison: Low Dose Pantoprazole (Approximately 0.3 mg/kg); Within group analysis of final week change from baseline for symptom Refusal to eat; Test type: Superiority or Other; p = 0.009, t-test, 2 sided
Statistical Analysis 6: Comparison: Low Dose Pantoprazole (Approximately 0.3 mg/kg); Within group analysis of final week change from baseline for symptom Difficulty swallowing; Test type: Superiority or Other; p = 0.004, t-test, 2 sided
Statistical Analysis 7: Comparison: High Dose Pantoprazole (Approximately 1.2 mg/kg); Within group analysis of final week change from baseline for symptom Difficulty swallowing; Test type: Superiority or Other; p = 0.044, t-test, 2 sided
Statistical Analysis 8: Comparison: Low Dose Pantoprazole (Approximately 0.3 mg/kg); Within group analysis of final week change from baseline for symptom Abdominal/belly pain; Test type: Superiority or Other; p = 0.002, t-test, 2 sided
Statistical Analysis 9: Comparison: Medium Dose Pantoprazole (Approximately 0.6 mg/kg); Within group analysis of final week change from baseline for symptom Abdominal/belly pain; Test type: Superiority or Other; p = 0.026, t-test, 2 sided
Statistical Analysis 10: Comparison: High Dose Pantoprazole (Approximately 1.2 mg/kg); Within group analysis of final week change from baseline for symptom Abdominal/belly pain; Test type: Superiority or Other; p = 0.026, t-test, 2 sided

3. Secondary Outcome: Change in Individual Weekly Mean Score For Each Respiratory Symptom From Baseline
Description: Individual respiratory symptoms weekly score was calculated as the average score / number of events for a patient in the corresponding week if the patient answered a question ≥3 times that week. Change = final week score minus baseline score. Final week was defined as the last 7 days of scores collected in the treatment period.
Time Frame: Baseline and 8 weeks
Population: The analysis population is all patients who were randomized and received ≥1 dose of test article and had nonerosive gastroesophageal reflux disease. Data were excluded if a patient answered a question <3 times in a week.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Low Dose Pantoprazole (Approximately 0.3 mg/kg) | Medium Dose Pantoprazole (Approximately 0.6 mg/kg) | High Dose Pantoprazole (Approximately 1.2 mg/kg)
Number analyzed (Participants) | 18 | 19 | 19
units on scale
  Presence of cold or fever: scale 1=yes 0=no | 0.11 (0.41) | 0.13 (0.43) | 0.11 (0.52)
  Cough without cold: scale 1=yes 0=no | -0.38 (0.34) | -0.20 (0.38) | -0.24 (0.36)
  Noisy breathing: scale 0(none)-3(most of the time) | -0.48 (0.97) | -0.19 (0.35) | -0.16 (0.36)
  Noisy breathing on exhale: scale 1=yes 0=no | -0.11 (0.55) | -0.15 (0.29) | -0.16 (0.29)
  Wheezing or whistling sound: scale 1=yes 0=no | -0.15 (0.46) | -0.04 (0.12) | -0.02 (0.08)
  Noisy breathing on inhale: scale 1=yes 0=no | -0.11 (0.49) | -0.16 (0.30) | -0.16 (0.31)
  Croupy or barky sound: scale 1=yes 0=no | -0.09 (0.30) | -0.03 (0.11) | -0.13 (0.32)
Statistical Analysis 1: Comparison: Low Dose Pantoprazole (Approximately 0.3 mg/kg); Within group analysis of final week change from baseline for Cough without cold; Test type: Superiority or Other; p = 0.004, t-test, 2 sided
Statistical Analysis 2: Comparison: Medium Dose Pantoprazole (Approximately 0.6 mg/kg); Within group analysis of final week change from baseline for Noisy breathing; Test type: Superiority or Other; p = 0.047, t-test, 2 sided

4. Secondary Outcome: Number of Patients With "Healed" Erosive Esophagitis (EE) at End of Study
Description: Healed EE was defined as a modified Hetzel-Dent (HD) score <2 on endoscopy at end of study. HD is a standardized rating scale for grading esophageal damage and severity of gastroesophageal reflux disease (GERD). HD score ranges from 0 (normal mucosa) to 4 (deep peptic ulceration).
Time Frame: 8 weeks
Population: The analysis population is randomized patients with erosive esophagitis at baseline.
Measure: Number; unit: patients
Arm/Group | Low Dose Pantoprazole (Approximately 0.3 mg/kg) | Medium Dose Pantoprazole (Approximately 0.6 mg/kg) | High Dose Pantoprazole (Approximately 1.2 mg/kg)
Number analyzed (Participants) | 0 | 2 | 2
patients | 0 | 2 | 2

ADVERSE EVENTS:
Arm/Group | Low Dose Pantoprazole (Approximately 0.3 mg/kg) | Medium Dose Pantoprazole (Approximately 0.6 mg/kg) | High Dose Pantoprazole (Approximately 1.2 mg/kg)
Serious Adverse Events (participants affected / at risk) | 0 | 1 | 1
Other Adverse Events (participants affected / at risk) | 18 | 19 | 18
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Low Dose Pantoprazole (Approximately 0.3 mg/kg) | Medium Dose Pantoprazole (Approximately 0.6 mg/kg) | High Dose Pantoprazole (Approximately 1.2 mg/kg)
Abdominal pain (General disorders) | 0/18 | 1/21 | 0/21
Anorexia (Gastrointestinal disorders) | 0/18 | 0/21 | 1/21
Dehydration (Metabolism and nutrition disorders) | 0/18 | 0/21 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Low Dose Pantoprazole (Approximately 0.3 mg/kg) | Medium Dose Pantoprazole (Approximately 0.6 mg/kg) | High Dose Pantoprazole (Approximately 1.2 mg/kg)
Abdominal pain (General disorders) | 1/18 | 1/21 | 3/21
Accidental injury (General disorders) | 3/18 | 3/21 | 2/21
Fever (General disorders) | 2/18 | 5/21 | 4/21
Flu syndrome (General disorders) | 0/18 | 1/21 | 1/21
Headache (General disorders) | 3/18 | 1/21 | 4/21
Infection (General disorders) | 1/18 | 0/21 | 1/21
Injection site hypersensitivity (General disorders) | 0/18 | 1/21 | 0/21
Lab test abnormal (General disorders) | 0/18 | 0/21 | 1/21
Pain (General disorders) | 1/18 | 0/21 | 0/21
Hemorrhage (Cardiac disorders) | 1/18 | 0/21 | 0/21
Anorexia (Gastrointestinal disorders) | 0/18 | 0/21 | 1/21
Constipation (Gastrointestinal disorders) | 1/18 | 0/21 | 1/21
Diarrhea (Gastrointestinal disorders) | 4/18 | 2/21 | 3/21
Gastroenteritis (Gastrointestinal disorders) | 1/18 | 1/21 | 2/21
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0/18 | 0/21 | 1/21
Gingivitis (Gastrointestinal disorders) | 0/18 | 0/21 | 1/21
Nausea (Gastrointestinal disorders) | 0/18 | 0/21 | 1/21
Rectal hemorrhage (Gastrointestinal disorders) | 0/18 | 0/21 | 1/21
Tooth cavities (Gastrointestinal disorders) | 1/18 | 0/21 | 0/21
Tooth disorder (Gastrointestinal disorders) | 1/18 | 1/21 | 0/21
Vomiting (Gastrointestinal disorders) | 2/18 | 4/21 | 3/21
Ecchymosis (Blood and lymphatic system disorders) | 2/18 | 1/21 | 1/21
Lymphadenopathy (Blood and lymphatic system disorders) | 1/18 | 1/21 | 3/21
Dehydration (Metabolism and nutrition disorders) | 0/18 | 1/21 | 1/21
Failure to thrive (Metabolism and nutrition disorders) | 0/18 | 1/21 | 0/21
Hyperlipemia (Blood and lymphatic system disorders) | 0/18 | 0/21 | 1/21
Peripheral edema (Metabolism and nutrition disorders) | 1/18 | 0/21 | 1/21
Ataxia (Nervous system disorders) | 0/18 | 0/21 | 1/21
Hyperkinesia (Nervous system disorders) | 0/18 | 0/21 | 1/21
Sleep disorder (Nervous system disorders) | 0/18 | 1/21 | 0/21
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/18 | 0/21 | 1/21
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0/18 | 0/21 | 1/21
Cough increased (Respiratory, thoracic and mediastinal disorders) | 3/18 | 3/21 | 1/21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/18 | 1/21 | 1/21
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0/18 | 1/21 | 1/21
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 3/18 | 2/21 | 0/21
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3/18 | 1/21 | 5/21
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1/18 | 0/21 | 2/21
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 8/18 | 7/21 | 8/21
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1/18 | 0/21 | 0/21
Contact dermatitis (Skin and subcutaneous tissue disorders) | 0/18 | 1/21 | 1/21
Exfoliative dermatitis (Skin and subcutaneous tissue disorders) | 0/18 | 0/21 | 1/21
Maculopapular rash (Skin and subcutaneous tissue disorders) | 0/18 | 0/21 | 1/21
Rash (Skin and subcutaneous tissue disorders) | 1/18 | 1/21 | 0/21
Urticaria (Skin and subcutaneous tissue disorders) | 0/18 | 1/21 | 0/21
Ear pain (Ear and labyrinth disorders) | 1/18 | 0/21 | 0/21
Eye pain (Eye disorders) | 1/18 | 0/21 | 0/21
Otitis media (Ear and labyrinth disorders) | 1/18 | 0/21 | 1/21
Urinary tract infection (Renal and urinary disorders) | 0/18 | 0/21 | 1/21
Vulvovaginal disorder (Reproductive system and breast disorders) | 1/18 | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.